CLINICAL TRIAL: NCT06147973
Title: Wellness Achieved Through Changing Habits (WATCH): An Acceptance-Based Healthy Lifestyle Intervention for Diverse Adolescents
Brief Title: An Acceptance-Based Healthy Lifestyle Intervention for Diverse Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Principal Investigator, Stephanie Manasse, Assistant Professor, Drexel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2306009959
Record Dates: First submitted 2023-11-10; First posted 2023-11-28 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Overweight and Obesity
Keywords: adolescent obesity; cardiovascular disease risk; healthy lifestyle intervention; acceptance-based
MeSH Terms: conditions — Overweight; Obesity; Pediatric Obesity | interventions — Helium

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either an acceptance-based treatment intervention or a health education comparison for the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance-based Treatment (ABT) (Experimental): ABT will consist of 18, 90-minute group sessions over 6 months.
  Interventions: Behavioral: Acceptance-based Treatment (ABT)
- Health Education (HE) Comparison (Sham Comparator): HE will include nine, 75-minute group health education sessions handouts over 6 months.
  Interventions: Behavioral: Health Education (HE) Comparison

INTERVENTIONS:
Behavioral: Acceptance-based Treatment (ABT) — Participants will be provided with psycho-education, skill-builders, and other coaching to promote weight loss and healthy lifestyle changes.
  Arms: Acceptance-based Treatment (ABT)
Behavioral: Health Education (HE) Comparison — Participants will be provided with psych-education and resources to promote weight loss and healthy lifestyle changes. They will not be provided with directives.
  Arms: Health Education (HE) Comparison

SUMMARY:
The goal of this clinical trial is to learn about cardiovascular disease risk among adolescent girls with overweight/obesity. The main questions this trial aims to answer are:

1. Does an acceptance-based healthy lifestyle intervention demonstrate more weight loss than a health education intervention?
2. Does an acceptance-based healthy lifestyle intervention show more improvements in participants' physiological, health-related, and psychological factors compared to a health education intervention?

Participants in this trial will:

1. Engage in treatment for 6-months, comprising of a mixture of in-person and remote group sessions, occurring at Drexel University or over a video-conferencing platform.
2. Complete various assessments. These include self-reported questionnaires, measures of weight, height, body composition, blood pressure, and blood lipids, and wearing of smart watches to measure sleep and physical activity.

Researchers will compare the acceptance-based and health education intervention groups to see if the acceptance-based treatment will indeed be effective in improving participants' health outcomes.

DETAILED DESCRIPTION:
Overweight/obesity (OW/OB) affects 14 million adolescents in the U.S. and disproportionately affects girls and racial/ethnic minorities while increasing their risk of cardiovascular disease (CVD) and type 2 diabetes. Adolescents demonstrate limited self-regulation skills, which are essential for adhering to diet and physical activity goals. Adolescents must contend with pervasive biological and environmental cues (e.g., cravings, labor-saving devices) that promote overeating and sedentary behavior. There is a critical need for interventions that teach self-regulation to enable adolescents to respond adaptively to these cues. Acceptance-based therapy (ABT) is an innovative approach that focuses on self-regulation skills, mindfulness, and increasing tolerance of uncomfortable internal experiences. There is strong evidence for ABT as an effective weight loss intervention for adults. The investigators conducted formative work using an adolescent-engaged approach to develop, implement, and feasibility test an ABT intervention for adolescent girls with OW/OB. The objective of this proposal is to test the efficacy of a novel ABT weight loss intervention tailored for adolescent girls with OW/OB.

This trial is the first to investigate ABT tailored for adolescent girls with OW/OB. The investigators will conduct a 6-month, randomized controlled trial comparing ABT with a health education comparison for 14- to 19-year-old adolescent girls with OW/OB, including ≥40% racial/ethnic minorities. To enhance scalability, interventions in both conditions will be delivered by bachelor's level paraprofessional weight loss coaches, treatment will occur in a hybrid of in-person and remote sessions, and the trial will take place in an outpatient community clinic. Assessments will be conducted at baseline, mid-treatment (month 3), post-treatment (month 6), 6-month follow-up (month 12), and 12-month follow-up (month 18), for a total study time of 18 months. The primary hypothesis is that adolescents randomized to ABT will exhibit significantly greater improvements in BMI z-score post-treatment compared to a health education comparison (HE). In the secondary aims, the investigators hypothesize that at post-treatment and 6- and 12-month follow-up, adolescents randomized to ABT will exhibit significantly greater improvements in their physiological, behavioral, and psychological risk factors compared to HE.

ELIGIBILITY:
Inclusion Criteria:

* Ages 14-19
* Gender identification as girl
* BMI percentile ≥ 85th percentile for sex-and-age

Exclusion Criteria:

* Experience of weight loss of ≥5% of body weight in the past 6 months for any reason except post-partum weight loss
* Having recently begun or changed the dosage of any medication known to affect appetite or body composition within the last 3 months
* Plans to move out of the area within the next year
* Active cancer or cancer requiring treatment in the past 2 years (except non-melanoma skin cancer)
* Active or chronic infections (e.g., HIV or TB)
* Active cardiovascular disease or event including hospitalization or therapeutic procedures for treatment of heart disease in the past 6 months
* Active kidney disease
* History of bariatric surgery
* Lung disease: chronic obstructive airway disease requiring use of oxygen (e.g., emphysema or chronic bronchitis)
* Diagnosed diabetes (type 1 or 2)
* Any condition prohibiting physical activity
* Diagnosis of an eating disorder
* Have a mental handicap or are currently experiencing other severe psychopathology that would limit their ability to engage in the treatment program (e.g., severe depression, active psychotic disorder)
* Recent or ongoing problem with drug abuse, alcohol abuse, or addiction
* Currently pregnant or less than 3 months post-partum
* Anticipation of a possible pregnancy in the next year
* Unwillingness to report possible or confirmed pregnancies promptly during the course of the trial

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — The participant must self-identify as female.
Enrollment: 148 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
BMI z-score change | Month 6
  Compare ABT vs. HE on BMI z-score change at post-treatment (month 6). The investigators hypothesize a significantly greater decrease in BMI z-scores in the ABT relative to HE.

SECONDARY OUTCOMES:
Physiological - Adiposity | Month 6, month 12, month 18
  Compare change in percent body fat in ABT relative to HE
Physiological - Blood pressure | Month 6, month 12, month 18
  Compare change in diastolic and systolic blood pressure in ABT relative to HE
Physiological - Blood lipids | Month 6, month 12, month 18
  Compare change in total blood lipid levels in ABT relative to HE. HDL, LDL, and total cholesterol will each be examined.
Health-related behaviors - dietary intake | Month 6, month 12, month 18
  Compare change in dietary intake in ABT relative to HE. Dietary intake will be measured with a VioScreen Food Frequency Questionnaire.
Health-related behaviors - physical activity | Month 6, month 12, month 18
  Compare change in physical activity in ABT relative to HE. Physical activity will be measured with a smart watch.
Psychological - Quality of life | Month 6, month 12, month 18
  Compare change in quality of life, in ABT relative to HE. Quality of life will be measured with the Quality of Life Inventory.
Psychological - Depression | Month 6, month 12, month 18
  Compare change in depression in ABT relative to HE at all time points. Depression will be measured using Beck's Depression Inventory-II.
Psychological - Disordered eating | Month 6, month 12, month 18
  Compare change in disordered eating in ABT relative to HE at all time points. Disordered eating will be measured using the Eating Disorder Examination Questionnaire.
Psychological - Psychological flexibility | Month 6, month 12, month 18
  Compare change in psychological flexibility in ABT relative to HE at all time points. Psychological flexibility will be measured using the Acceptance and Action Questionnaire II.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Manasse, PhD, Principal Investigator — Drexel University
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with the study Data Safety Monitoring Board (DSMB). Following study close-out, de-identified data and related data dictionaries will be available upon request.
Time Frame: Data will be available upon request following the conclusion of the study.
Access Criteria: For access, interested parties must contact the principal investigator.

REFERENCES:
- [Background] Ogden CL, Carroll MD, Lawman HG, Fryar CD, Kruszon-Moran D, Kit BK, Flegal KM. Trends in Obesity Prevalence Among Children and Adolescents in the United States, 1988-1994 Through 2013-2014. JAMA. 2016 Jun 7;315(21):2292-9. doi: 10.1001/jama.2016.6361. PMID 27272581
- [Background] Newsome FA, Cardel MI, Chi X, Lee AM, Miller D, Menon S, Janicke DM, Gurka MJ, Butryn ML, Manasse S. Wellness Achieved Through Changing Habits: A Randomized Controlled Trial of an Acceptance-Based Intervention for Adolescent Girls With Overweight or Obesity. Child Obes. 2023 Dec;19(8):525-534. doi: 10.1089/chi.2022.0116. Epub 2022 Nov 17. PMID 36394498